CLINICAL TRIAL: NCT00768625
Title: Cardiovascular Risk Stratification in Patients With Obstructive Sleep Apnea
Acronym: ERA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Responsible Party: Fatima Dumas Cintra, AFIP
Other Study IDs: ERA
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is:

1. To determine the frequency of cardiovascular diseases in patients with OSA, obese, overweight, and lean (BMI<25)
2. To analyze the CPAP treatment over the clinical evolution of OSA patients
3. To determine if OSA is a independent predictor of cardiovascular risk

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a condition with important cardiovascular repercussions. However, the association between OSA, cardiovascular diseases, and obesity has not been totally clarified. We hypothesized that the cardiovascular consequences of OSA are due to obesity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with OSA (apnea-hypopnea index higher than 5 events/hour)

Exclusion Criteria:

* Body mass index higher than 40

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 OSA patients and 1000 controls enrolled from Instituto do Sono database 500 subjects with body mass index less than 25
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-04; Primary Completion 2011-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | five years

CONTACTS AND LOCATIONS:
Overall Officials: Fatima D Cintra, PhD, Principal Investigator — Associacao Fundo de Incentivo a Psicofarmcologia; Dalva Poyares, PhD, Study Chair — Associacao Fundo de Incentivo a Psicofarmcologia; Sergio Tufik, PhD, Study Director — Associacao Fundo de Incentivo a Psicofarmcologia
Locations (1):
- Instituto do Sono/AFIP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Feres MC, Fonseca FA, Cintra FD, Mello-Fujita L, de Souza AL, De Martino MC, Tufik S, Poyares D. An assessment of oxidized LDL in the lipid profiles of patients with obstructive sleep apnea and its association with both hypertension and dyslipidemia, and the impact of treatment with CPAP. Atherosclerosis. 2015 Aug;241(2):342-9. doi: 10.1016/j.atherosclerosis.2015.05.008. Epub 2015 May 23. PMID 26071656
- [Derived] Cintra FD, Tufik S, Paola Ad, Feres MC, Melo-Fujita L, Oliveira W, Rizzi C, Poyares D. Cardiovascular profile in patients with obstructive sleep apnea. Arq Bras Cardiol. 2011 Apr;96(4):293-9. doi: 10.1590/s0066-782x2011005000030. Epub 2011 Mar 18. English, Portuguese, Spanish. PMID 21437515
- [Derived] Rizzi CF, Cintra F, Risso T, Pulz C, Tufik S, de Paola A, Poyares D. Exercise capacity and obstructive sleep apnea in lean subjects. Chest. 2010 Jan;137(1):109-14. doi: 10.1378/chest.09-1201. Epub 2009 Oct 3. PMID 19801583